CLINICAL TRIAL: NCT05341284
Title: Impact of HPV Vaccination on HPV Infection and Cervical Related Disease Burden in Real-World Settings (HPV-RWS): A Prospective Cohort
Brief Title: Impact of HPV Vaccination on HPV Infection and Cervical Related Disease Burden in Real-World Settings (HPV-RWS)
Acronym: HPV-RWS
Status: Withdrawn | Type: Observational
Why Stopped: Due to on-site coordination issues and lack of cooperation from the research site staff, the study was withdrawn.
Sponsor: Peking University (Other)
Collaborators: Center for Disease Control and Prevention of Yinzhou District, Ningbo City, China (Unknown); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: HPV-RWS
Record Dates: First submitted 2022-03-29; First posted 2022-04-22 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2022-04

CONDITIONS: HPV Infection; Cervical Disease
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: The subject who is receiving first or second dose of the AS04 adjuvanted HPV 16/18 vaccine at the enrollment.
  Interventions: Other: Questionnaire Survey and Cervical Cancer Screening
- Non-exposed group: The subject who does not have any HPV vaccination history at the enrollment or during the study period.
  Interventions: Other: Questionnaire Survey and Cervical Cancer Screening

INTERVENTIONS:
Other: Questionnaire Survey and Cervical Cancer Screening — A brief questionnaire will be administered to all participants at enrollment and at the pre-scheduled follow-up visit at Month 36.
  For the subject who are eligible for the screening (i.e. (1)≥ 18 years old; (2) had sexual debut prior to enrollment, (3) no contradiction to the screening, (4) voluntary to the screening) will be referred to the study site hospitals by offering the subjects a cervical cancer screening voucher, and the type-specific HPV test will be performed as primary screening approach at Month 0 and 36.

SUMMARY:
Take AS04 adjuvanted HPV16/18 vaccine as an example to evaluate the impact of HPV vaccination on HPV infection and related disease burden in the real world based on prospective cohort and Yinzhou Regional Health Information Platform (YRHIP), in order to bridge the gap in relevant evidence in China.

ELIGIBILITY:
Inclusion Criteria:

* Permanent female resident in the Yinzhou District (i.e. at least residing in the Yinzhou District for a 3-year period and at least 6months in every 12-month period).
* Between 9 and 45 years old at time of the enrollment.
* Receiving first or second dose of the AS04 adjuvanted HPV 16/18 vaccine (exposed group). Or without any HPV vaccination history (non-exposed group).
* Subjects and their parents / legal guardians agreed to comply with the requirements mentioned in the protocol (e.g., physically and mentally healthy, be able to complete the baseline and follow-up survey and would comply with the visits, etc.).
* Written informed consent will be obtained from the subject. For subjects who are below the legal age of consent, written informed consent must be obtained from the parent(s)/LAR(s) of the subject and informed assent must be obtained from the subject according to EC requirement as well as local law. Subjects must understand the protocol and be voluntarily willing to join this study with written informed consent form.

Exclusion Criteria:

* Pregnancy at the enrollment.
* Females with historical cervical diseases (i.e., CIN1, CIN2, CIN3, and cervical cancer) before the recruitment.
* After hysterectomy.
* Females with malignant tumor history or other severe diseases (e.g., liver failure, heart failure, etc.) whose life expectancy is less than 12 months.
* Females who (1) have historical HPV vaccination, or (2) are in non-exposed groups but have clear intention for HPV vaccination in next 3 years.

Ages: 9 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study will enroll the permanent female residents between 9 to 45 years old in the Yinzhou District, with AS04 adjuvanted HPV 16/18 vaccination history or without any HPV vaccination history.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Cervical infection with HPV-16 and/or HPV-18 (by PCR) | up to 36 month
  HPV-16 and/or HPV-18 infection is defined as at least one positive HPV-16 or HPV-18 DNA PCR assay at enrollment (Month 0) or follow-up (Month 36) or any additional screenings during the study period.

SECONDARY OUTCOMES:
The occurrence of high-risk HPV infection 12 other hr-HPV positive besides of type 16/18 | up to 36 month
  12 other hr-HPV positive besides of type 16/18 infection is defined as at least one positive for HPV 31/33/35/39/45/51/52/56/58/59/66/68 or multiple types DNA PCR assay at enrollment (Month 0) or follow-up (Month 36) or any additional screenings during the study period.
Number of Participants with Any cervical lesions or diseases | up to 36 month
  Any cervical lesions or diseases is defined as atypical squamous cells of undefined significance (ASC-US), atypical glandular cells (AGC), atypical squamous cells, cannot exclude for highly squamous intraepithelial lesions (ASC-H), low-grade squamous intraepithelial lesion (LSIL), high-grade squamous intraepithelial lesion (HSIL), Cervical Intraepithelial Neoplasia (CIN) 1, CIN2, CIN3, squamous cell carcinoma (SCC), adenocarcinoma in situ (AIS) and adenocarcinoma (ADC). Any hr-HPV type infection is defined as at least one positive for HPV 16/18/31/33/35/39/45/51/52/56/58/59/66/68 or multiple types DNA PCR assay in the aforesaid cervical sample.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Z, Li P, Zeng X, Yao X, Sun Y, Lin H, Shen P, Sun F, Zhan S. Impact of HPV vaccination on HPV infection and cervical related disease burden in real-world settings (HPV-RWS): protocol of a prospective cohort. BMC Public Health. 2022 Nov 18;22(1):2117. doi: 10.1186/s12889-022-14474-1. PMID 36401179